CLINICAL TRIAL: NCT05813210
Title: Myocardial Ischemia Detection With a Combined Cardiovascular Magnetic Resonance and Biomarker Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Olten (Other)
Responsible Party: Principal Investigator, Nisha Arenja, PD Dr. med. Nisha Arenja Leitende Ärztin, Department of Cardiology, Kantonsspital Olten, Solothurner Spitäler AG Baslerstrasse 150, 4600 Olten, Switzerland, Kantonsspital Olten
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ischemia-CMR-Biomarker
Record Dates: First submitted 2023-03-21; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Ischemia Demand
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, two-arm controlled, monocentric, national study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined stress test (pharmacological and physical stress) (Experimental): Patients are first stressed ergometrically and perfusion is assessed. Subsequently, drug induced stress perfusion is performed, as in the usual protocol.
  Interventions: Diagnostic Test: Exercise in combination with biomarkers and pharmacological stress CMR test
- Pharmacological stress test (Active Comparator): One group receiving only pharmacological stress test with Regadenoson.
  Interventions: Diagnostic Test: Exercise in combination with biomarkers and pharmacological stress CMR test

INTERVENTIONS:
Diagnostic Test: Exercise in combination with biomarkers and pharmacological stress CMR test — A bicycle ergometry combined with pharmacoligical stress test is performed. High sensitive Troponin is taken before and after the stress test.

SUMMARY:
Background:

Early detection and treatment of coronary artery disease (CAD) can help curb the high incidence of cardiovascular disease, which is the leading cause of death worldwide. Today, we have sophisticated imaging techniques available to diagnose CAD, including cardiovascular magnetic resonance (CMR). CMR is able to detect relevant myocardial ischemia and guide treatment options. Therefore, it is recommended by the current guidelines for patients at intermediate risk. In clinical practice, we often encounter two main issues: first, because of their availability and increasing uncertainty in the population, imaging techniques are increasingly used, even in patients with a low pretest probability for the presence of CAD. Second, the diagnostic accuracy of the techniques is not perfect, and false-negative stress CMR perfusion studies are an important limitation of the method, especially in patients with advanced CAD and balanced ischemia. In addition, the standard method with pharmacologic testing carries an inherent risk.

Aim:

The aim of our project is to review the clinical pretest probability to reduce unnecessary imaging studies and to evaluate the improvement of diagnostic accuracy of CMR stress testing by adding exercise test and reviewing biomarkers, which could reduce the number of false-negative results, especially in patients with balanced ischemia, who usually suffer from severe CAD.

Methodology:

This is a prospective, randomized, two-arm, controlled, monocentric, national study performed in collaboration by two centers (Solothurner Spitäler AG and CRIB). Included are consecutive patients with suspected inducible myocardial ischemia who are examined by CMR at the Kantonsspital Olten and during the course also at the Bürgerspital Solothurn. Since all patients from the Kanton Solothurn are referred to us for CMR diagnosis, this represents an ideal referral pattern of unselected patients with a wide range of pretest probability for myocardial ischemia (interquartile range of pretest probability 20-60%). Patients able to exercise will randomized to either standard CMR stress protocol with regadenoson or to the combined CMR stress protocol, which includes additional exercise testing and measurement of hs-cTn, a biomarker for detecting myocardial damage. Patients with positive CMR results will be received to coronary angiogram.

Potential Significance:

This project has the potential to reduce the residual risk and thereby reduce cardiovascular mortality in patients with false-negative test result, especially those with balanced ischemia or inadequate response to vasodilatation drugs. In addition, the investigator will be able to make a statement about the additional use of biomarkers for the diagnosis of CAD in patients with stable condition. Thereby, the integrated use of biomarkers may improve the diagnostic accuracy and this might prevent unnecessary further strategies, which will reduce high-cost in health care systems. Furthermore, the investigator hopse for better patient selection in order to avoid unnecessary examinations in the future.

DETAILED DESCRIPTION:
Study Category and Rationale: This test falls into risk category A, since the medical device bears a conformity mark and is handled in clinical practice over a long period of time in accordance with the instructions for use. The drugs have also been in use in clinical routine for years.

Background and Rationale: For the diagnosis of CAD, we currently dispose sophisticated imaging techniques including cardiovascular magnetic resonance (CMR). In clinical routine, we often encounter the following issues: First, because of their availability and increasing uncertainty in the population, imaging modalities are increasingly used, even in patients with a low pretest probability for the presence of CAD, which is associated with high costs. Second, the diagnostic accuracy of the techniques is neither perfect nor equivalent between modalities, and there is an inherent testing risk.

Risk / Benefit Assessment: The benefit/risk relationship for our patients is high, as there is no specific study related risks. The risk of a study includes the risks of the trial intervention itself (CMR stress testing and insertion of a venous access with blood collections) as well as the risk of unauthorized data access through third parties or unwanted identification of participants. The benefit of this study may be an improvement in CMR stress testing for better diagnostic accuracy so that relevant ischemia is not missed or patients do not undergo coronary angiography unnecessarily.

Primary endpoint:

MR combined stress test vs CMR standard stress test protocol. As a primary analysis, we will compare the relative number of positive cases of CAD identified by the CMR test (number of patients positive on CMR and consecutive positive on angiography as a proportion of the total number of patients in the randomization group).

Secondary endpoints:

* Patients tolerance of the test using modified Glasgow comfort score.
* Number of rehospitalisation, cardiac interventions, acute myocardial infarction and death in both CMR stress protocols after 12 months of follow-up.

Study Design: Prospective, randomized, two-arm controlled, monocentric, national study.

Statistical Considerations: The full analysis data set (FAS) consists of all patients who signed the informed consent and underwent the CMR stress test as described for the group Primary analysis As a primary analysis, the investigator will compare the relative number of positive cases of CAD identified by the CMR test (number of patients positive on CMR and consecutive positive on angiography as a proportion of the total number of patients in the randomization group). The investigator will compare these proportions using a chi-squared test. Assuming an equal prevalence of CAD in each group, due to the randomization taking risk factors into account as stratification factors, a difference in the proportion of true positive cases compared to angiography, will mean that there is a difference in sensitivity of the screening protocol.

Secondary analyses

The following secondary endpoints will be evaluated:

1. Feasibility of CMR exercise stress testing in clinical routine
2. Verification of the clinical pre-test probability on the basis of the assessment by the attending physician and hs-cTn.
3. Incidence of rehospitalisation, cardiac interventions, acute myocardial infarction and death in both CMR stress protocols after 12 months of follow-up.
4. Differences between exercise and pharmacological CMR perfusion scans.

The first secondary endpoint will be assessed descriptively using a patient-reported and physician- reported outcomes.

For investigate the second secondary objective, the investigator will describe the number of positive cases on angiography found by the physician's assessment and hs-cTn, respectively in each of the groups (hs-cTn only in the intervention group). The investigator will compare the number to the full stress test protocol within each group by a chi-squared test.

As a final secondary analysis, the investigator will assess the association between the CMR test result and group (with addition of the interaction between the two variables) and the time to the following outcome events:

* Rehospitalisation
* Cardiac intervention
* Acute myocardial infarction
* Death due to cardiovascular reasons
* Death due to any cause

The investigator will use Cox proportional hazard models to investigate if there is an association between the time to each of the abovementioned events, adn tha CMR test result and group allocation. Covariates that need to be added to these models will be assessed at a later stage.

Rational of sample size is explained below.

Number of Participants with Rationale: The sample size was determined using a resampling method to be able to show a difference in the proportion of patients with CAD on angiography in the two groups. The investigator evaluated different sample sizes and each sample size, ni=1,...,131 = 350, ..., 1000, was evaluated by simulating R = 10000 times ni individual patients. The simulated data sets had the following characteristics, based on available literature:

* Patients are randomized 1:1 to the two different groups
* In the control group, 20% of the patients has an indication of ischemia in the screening test and underwent angiography.
* The positive predictive value for both groups was assumed to be equal at 92%.
* In the intervention group the proportion of patients with an indication of ischemia was assumed to be 30%. This means that the investigator assumed that the addition of the two additional tests resulted in 10% more patients with an indication of ischemia during the screening.

In each simulated data set, the investigator compared the proportion of true positives (i.e. patients with indication of ischemia on the screening test and positive angiography) in the total group between the two groups using a Chi-squared test. The p-value was derived for each model to assess if there was a difference in proportion between the two groups. The investigator set the type I error probability, α, to 0.05, and examined the effect of type II error probabilities, β, 0.20 and 0.10 on the sample size. The null hypothesis, no difference between the two groups, was rejected if the p-value of the Chi-squared test was lower than α.

Figure 6 shows how the sample size depends on the prevalence of positive screening tests in the intervention group, with a probability of a positive screening test of 20% in the control group and a positive predictive value (PPV) of 92% in both groups. With an estimated drop out of 10 %, a total of 772 patients should be recruited to allow us with a power of 80% (i.e. in 80 out of 100 simulated studies) and a significance level of 0.05 (α) to show a difference in the proportion of true positives between the two groups.

Study Interventions: All patients, who will be sent to CMR for evaluation of hemodynamic relevant myocardial ischemia and who are able to exercise will be randomised either to the CMR standard stress using Regadenoson or to the CMR combined stress protocol using exercise and Regadenoson stress in combination with hs-cTn measurements.

Study Duration: The study inclusion is planned for 2 year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with suspected hemodynamic relevant myocardial ischemia with or without known CAD
* Patients able to give informed consent as documented by signature
* Patients able to physically able to exercise

Exclusion Criteria:

* Patients with acute coronary syndrome (ACS)
* Inability to exerciseInability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Contraindications to CMR implantable devices, cerebral aneurysm clips, cochlear implants
* Severe Claustrophobia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of positive cases of coronary artery disease using CMR combined stress test vs CMR standard stress test protocol. | 2 years
  Coronary angiography is performed in patients with positive CMR results of both groups.

SECONDARY OUTCOMES:
Patients tolerance of the test using modified Glasgow comfort score. | 1 year
  GCM descriptor: No: No discomfort, resting comfortably throughout, minimal: one or two episodes of mild discomfort, well tolerated, mild: more than two episodes of discomfort, adequately tolerated, moderate: significant discomfort, experienced several times throughout the procedure
Number of rehospitalisation, cardiac interventions, acute myocardial infarction and death in both CMR stress protocols after 12 months of follow-up. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Olten, Olten, Switzerland